CLINICAL TRIAL: NCT00418782
Title: A 2 Week, Randomized, Double Blind, Placebo And Positive Controlled, Parallel Group, Multicenter Study Of CE-224,535 In Subjects With Osteoarthritic Pain Of The Knee
Brief Title: A Study Of The Effect Of CE-224535 On Knee OA (Osteoarthritis) Pain
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Results of interim analysis indicate lack of efficacy when compared to placebo.
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A6341008
Record Dates: First submitted 2007-01-04; First posted 2007-01-05 (Estimated); Last update posted 2018-12-05 (Actual); Status verified 2018-12

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Naproxen; CE 224,535

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator)
  Interventions: Drug: naproxen
- 2 (Experimental)
  Interventions: Drug: CE-224535
- 3 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: naproxen
  Arms: 1
Drug: CE-224535
  Arms: 2
Drug: placebo
  Arms: 3

SUMMARY:
CE-224535 is a new medication being developed as an analgesic and anti-inflammatory agent for the treatment of the signs and symptoms of osteoarthritis (OA). The purpose of this study is to evaluate the analgesic and anti inflammatory efficacy and safety of CE 224,535 versus placebo and naproxen treatment in patients with OA knee pain.

ELIGIBILITY:
Inclusion Criteria:

* Is a healthy adult 18 to 75 years of age, inclusive, in general good health and with diagnosis of knee OA, as determined by the American College of Rheumatology (ACR) clinical/radiographic classification criteria for OA of the knee.
* Women must be of non childbearing potential (amenorrhea for at least 1 year PLUS have a serum follicle stimulating hormone (FSH) level >30 IU/L, bilateral oophorectomy or hysterectomy), and have a confirmed negative serum pregnancy test at the screening visit prior to randomization.

Exclusion Criteria:

* History of other diseases that may involve the study joint, including inflammatory joint diseases, crystalline disease, endocrinopathies, metabolic diseases, infections, neuropathic disorders, avascular necrosis, Paget's disease, or tumors.
* Women of childbearing potential, or who are pregnant or lactating.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2007-01; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
To determine the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of oral multiple doses of CE 224,535 in subjects with OA of the knee | ongoing
The primary endpoint is the change from Baseline (Day 1) to Week 2 (Day 14) in the WOMAC Pain domain score. | Day 1-14

SECONDARY OUTCOMES:
The change from Baseline to each day (Days 1 to 6) and over the average response in Days 1 to 6 using an 11 point numeric rating scale (NRS) from 0-10 on daily pain diary; | (Days 1 to 6)
Patient's Global Impression of Change (PGIC) at Week 2; | Week 2
The change from Baseline to Weeks 1 and 2 in the Patient's Global Assessment of Arthritic Condition; | Baseline to Weeks 1 and 2
The change from Baseline to Week 1 (Day 7) in the WOMAC Pain domain score; | Day 7
The change from Baseline to Weeks 1 and 2 (Days 7 and 14) in the WOMAC Stiffness domain score; | Days 7 and 14
The change from Baseline to Weeks 1 and 2 (Days 7 and 14) in the WOMAC Physical Function domain score; | Days 7 and 14
The change from Baseline to Weeks 1 and 2 (Days 7 and 14) in the WOMAC Total Score by simple summation; | Days 7 and 14
The change from Baseline to Weeks 1 and 2 (Days 7 and 14) in the WOMAC Importance Weighted Total Score; | Days 7 and 14
The change from Baseline to Weeks 1 and 2 in the Patient's Assessment of Arthritis Pain (VAS) | Weeks 1 and 2

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (42):
- United States (42):
  - Pfizer Investigational Site, Anniston, Alabama
  - Pfizer Investigational Site, Bayou La Batre, Alabama
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, Hot Springs, Arkansas
  - Pfizer Investigational Site, Northridge, California
  - Pfizer Investigational Site, Sacramento, California
  - Pfizer Investigational Site, Tarzana, California
  - Pfizer Investigational Site, Denver, Colorado
  - Pfizer Investigational Site, Westminster, Colorado
  - Pfizer Investigational Site, Clearwater, Florida
  - Pfizer Investigational Site, DeFuniak Springs, Florida
  - Pfizer Investigational Site, Destin, Florida
  - Pfizer Investigational Site, Pensacola, Florida
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Gurnee, Illinois
  - Pfizer Investigational Site, Avon, Indiana
  - Pfizer Investigational Site, Indianapolis, Indiana
  - Pfizer Investigational Site, Gretna, Louisiana
  - Pfizer Investigational Site, Kenner, Louisiana
  - Pfizer Investigational Site, Metairie, Louisiana
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Frederick, Maryland
  - Pfizer Investigational Site, Flowood, Mississippi
  - Pfizer Investigational Site, Columbia, Missouri
  - Pfizer Investigational Site, Kansas City, Missouri
  - Pfizer Investigational Site, Missoula, Montana
  - Pfizer Investigational Site, Trenton, New Jersey
  - Pfizer Investigational Site, Beavercreek, Ohio
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Kettering, Ohio
  - Pfizer Investigational Site, Ashland, Oregon
  - Pfizer Investigational Site, Eugene, Oregon
  - Pfizer Investigational Site, Duncansville, Pennsylvania
  - Pfizer Investigational Site, Summerville, South Carolina
  - Pfizer Investigational Site, Collierville, Tennessee
  - Pfizer Investigational Site, Knoxville, Tennessee
  - Pfizer Investigational Site, Memphis, Tennessee
  - Pfizer Investigational Site, Bryan, Texas
  - Pfizer Investigational Site, Longview, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Arlington, Virginia
  - Pfizer Investigational Site, Spokane, Washington

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6341008&StudyName=A%20Study%20Of%20The%20Effect%20Of%20CE-224535%20On%20Knee%20OA%20%28Osteoarthritis%29%20Pain